CLINICAL TRIAL: NCT05385133
Title: Condyle Repositioning Using Patient Specific Guides and Prebent Plates Osteosynthesis Versus Conventional Mandibular Bilateral Sagittal Split Osteotomy Set-back Surgery: A Randomized Clinical Trial
Brief Title: Condyle Repositioning Using PSI and Prebent Plates Osteosynthesis Versus Conventional Mandibular BSSO Set-back Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Ali, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMFS-14719
Record Dates: First submitted 2022-05-07; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Orthognathic Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer guided condylar position (Experimental): post-osteotomy condylar position was performed using patient specific surgical guides and pre-bent plates
  Interventions: Procedure: Computer guided condylar position
- Manual condylar position (Experimental): post-osteotomy condylar position was performed using the conventional free hand approach
  Interventions: Procedure: Manual condylar position

INTERVENTIONS:
Procedure: Computer guided condylar position — post-osteotomy condylar position was performed using patient specific surgical guides and pre-bent plates
  Arms: Computer guided condylar position
Procedure: Manual condylar position — post-osteotomy condylar position was performed using the conventional manual method
  Arms: Manual condylar position

SUMMARY:
Patients with skeletal class III malocclusion were allocated to two groups. Both proximal and distal segments were repositioned using osteotomy/screw holes and plate locating surgical guides with pre-bent plates osteosynthesis in the intervention group, while manual free hand condylar segment seating was used for proximal segment positioning in the control group.

DETAILED DESCRIPTION:
Twenty patients with skeletal class III malocclusion were randomly allocated to two groups. Both proximal and distal segments were repositioned using osteotomy/screw holes and plate locating surgical guides with pre-bent plates osteosynthesis in the intervention group, while manual free hand condylar segment seating was used for proximal segment positioning in the control group. Accuracy of condylar position was assessed using computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients complaining of skeletal class III malocclusion that require BSSO for correction of their deformity

Exclusion Criteria:

* Patients require bi-maxillary orthognathic surgery
* patients with temporomandibular joint dysfunction

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Condylar deviation | 1 week postoperatively
  Change of condyle position postoperative from preoperative position

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No